CLINICAL TRIAL: NCT03275792
Title: Inpatient Volume Expansion in Children With Shiga Toxin-Producing Escherichia Coli (STEC) Infection to Prevent Hemolytic Uremic Syndrome (HUS)
Brief Title: Shiga Toxin Producing Escherichia Coli (STEC) Volume Expansion
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding not obtained.
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHREB-12345
Record Dates: First submitted 2017-08-29; First posted 2017-09-08 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2019-09

CONDITIONS: Hemolytic-Uremic Syndrome
Keywords: Shiga-Toxigenic Escherichia coli; Child
MeSH Terms: conditions — Hemolytic-Uremic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Admission/Intravascular Volume Expansion (Experimental): 1. Infusion of 40 mL/kg of 0.9% normal saline (NS) IV over 60 minutes
  2. 0.9% NS with 5% dextrose at 150% of standard maintenance volume
  3. If urine output is <0.5 ml/kg/hr over a 12-hour period (AKI Stage 2), repeat 20 mL/kg bolus or boluses of 0.9% NS will be infused as long as there are no signs of central volume overload
  4. Oral fluids ad lib along with strict input/output documentation
  5. Fluids will be restricted if: A) Anuria for 12 hours OR B) Evidence of fluid overload
  6. Daily laboratory tests and in-person assessment until inpatient discharge criteria reached:
     A) 2 - 4 days since symptom onset AND rising platelet count (>5% increase) documented over 48 hours in a clinically well child B) ≥5 days since symptom onset AND stable platelet count (<5% decrease) documented over 48 hours in a clinically well child
  7. Repeat hematocrit, platelet, renal function 24 and 72-hours post-discharge.
  Interventions: Drug: D5-0.9%NS
- Outpatient Observation (Active Comparator): 1. Following standard emergency department (ED) care [volume status assessed; dehydration corrected employing oral rehydration in children with mild to moderate dehydration (most common); IV if severe (rarely)], children are discharged with saline lock IV (routine procedure across Canadian pediatric EDs).
  2. Oral fluids (preferably electrolyte maintenance solutions) ad lib following ED discharge
  3. Additional health assessments as required
  4. Daily blood tests at a local laboratory with results conveyed daily to the site-investigator until outpatient discharge criteria achieved; no in-person assessment given logistics (i.e. distance), impact on family, and mirroring of standard practice A) 2 - 4 days since symptom onset AND rising platelet count (>5% increase) documented over 48 hours in a clinically well child B) ≥5 days since symptom onset AND stable platelet count (<5% decrease) documented over 48 hours in a clinically well child
  Interventions: Drug: Routine home oral rehydration

INTERVENTIONS:
Drug: D5-0.9%NS — Admission for intravascular volume expansion
  Arms: Admission/Intravascular Volume Expansion
Drug: Routine home oral rehydration — Routine oral fluids as is given at home to all children with acute diarrheal disease
  Arms: Outpatient Observation

SUMMARY:
This study will provide feasibility data regarding the conduct of a clinical trail evaluating the use of early aggressive inpatient intravenous rehydration in children with Shiga Toxin producing E. coli infection.

DETAILED DESCRIPTION:
Background: Shiga toxin-producing Escherichia coli (STEC) cause a spectrum of disease, ranging from asymptomatic carriage to bloody diarrhea and the hemolytic uremic syndrome (HUS). HUS is caused by a toxin that destroys red blood cells, consumes platelets and impairs kidney function. HUS results in morbidity and even death in otherwise healthy children. Over the last 30 years however, there has been extremely limited progress in preventing acute and long-term complications in children with STEC infection. However, it is believed that Shiga toxins generate clots or blockages in the kidneys that damage it much the way strokes cause brain damage. There is emerging evidence that if children with STEC infection are recognized early, then the interval between diarrhea onset and the presence of HUS could be exploited to preserve kidney function through the use of intravenous rehydration.

Study Design: The investigators propose to conduct the first randomized clinical trial of volume expansion therapy in children with STEC infection. Employing Alberta's unique province-wide microbiology network and its only two pediatric tertiary care centres, the investigators will conduct a proof of principal feasibility study that evaluates novel technologies to identify STEC infected children and those at risk for HUS.

Objectives: The primary outcome will be process: number of children recruited. Secondary outcomes will include: 1) resources: retention; refusal; compliance; eligibility criteria; questionnaires; data collection tools; and time requirements; 2) management: capacity and impact on clinical services; 3) scientific: utility of point-of-care STEC diagnostics; use of urine biomarkers to identify high risk children, monitoring of kidney injury and response to therapy; and safety.

Significance: This pilot will provide the necessary data to integrate novel technologies into the design and conduct of a multicentre, multinational, clinical trial that will reduce morbidity and mortality from STEC infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age <18.0 years;
2. STEC infection [positive culture OR antigen OR polymerase chain reaction test for Stx/gene];
3. Day of illness 1-10: Children who develop HUS will do so by day #14 of illness;8 restricting enrolment to the first 10 days will ensure all participants are at risk of HUS.

Exclusion Criteria:

1. Evidence of evolving HUS: A) Hematocrit <30% OR B) Platelet count <150 x 109/L;
2. Responsible physician desires patient admission (therefore unable to randomize);
3. Unable to contact family within 48 hours of positive stool test;
4. Patient with history of atypical HUS;
5. Chronic disease limiting fluid volumes administered (e.g. impaired cardiac function)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Number of children enrolled in the study protocol | at the end of the 24 month study recruiting period
  The number of children recruited per month per site will be calculated and will be related to the number screened, number eligible, and number consented.

SECONDARY OUTCOMES:
The proportion of children enrolled in each study arm who develop adverse events | at the end of the 24 month study recruiting period
  For participants enrolled in each study arm we will quantify the proportion that are admitted to Intensive Care Units, the proportion requiring respiratory support (CPAP, BiPAP, endotracheal intubation), hypoxia defined by the administration of supplemental oxygen, and evidence of congestive heart failure defined by blinded independent reviewers.
Retention | at the end of the 24 month study recruiting period
  The proportion of children who complete the study protocol
Time requirements | at the end of the 24 month study recruiting period
  We will quantify the number of hours children remain admitted and to which clinical units
Child/family perspectives | at the end of the 24 month study recruiting period
  7-item likert scales will be employed to evaluate perspectives of parents and participants as appropriate related to study protocols, procedures and participation
compliance/adherence | at the end of the 24 month study recruiting period
  The proportion of children enrolled in each study arm who comply with the key interventions of the respective study arms
data collection tool performance | at the end of the 24 month study recruiting period
  Individual data fields will be audited with respect to data quality, reliability, completeness, timeliness of completion
Impact on clinical services | at the end of the 24 month study recruiting period
  We will qualitatively explore with the department leads at the respective institutions if the study protocol had any impact on clinical care provided either to the admitted patients or to other patients on their services
Cost | at the end of the 24 month study recruiting period
  We will quantify the costs per child in each study arm

OTHER OUTCOMES:
Point-of-Care STEC diagnosis | at the end of the 24 month study recruiting period
  diagnostic accuracy compared with standard culture
Urine biomarkers | at the end of the 24 month study recruiting period
  ability to predict progression to AKI and HUS
Point-of-Care STEC diagnosis | at the end of the 24 month study recruiting period
  turnaround time
Point-of-Care STEC diagnosis | at the end of the 24 month study recruiting period
  proportion O157 vs other STEC

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MDCM, MSc, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Imdad A, Mackoff SP, Urciuoli DM, Syed T, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD012997. doi: 10.1002/14651858.CD012997.pub2. PMID 34219224